CLINICAL TRIAL: NCT07223424
Title: Patient Preference for Subcutaneous vs. Intravenous Immune Therapy (PSI-Immune)
Brief Title: Patient Preference for Subcutaneous vs. Intravenous Immune Therapy
Acronym: PSI-Immune
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HCC 25-125
Record Dates: First submitted 2025-10-23; First posted 2025-10-31 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Renal Cell Carcinoma; Non Small Cell Lung Cancer; Melanoma; Colo-rectal Cancer (dMMR/MSI-H CRC); Hepatocellular Carcinoma; Ulcerative Colitis; Esophageal Cancer; Squamous Cell Carcinoma; Gastric/GEJ; Cervical Cancer; Gastro-Esophageal Adenocarcinoma; Esophageal Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Melanoma; Colonic Neoplasms; Carcinoma, Hepatocellular; Colitis, Ulcerative; Esophageal Neoplasms; Carcinoma, Squamous Cell; Uterine Cervical Neoplasms; Adenocarcinoma Of Esophagus | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subcutaneous to IV (Active Comparator): SC nivolumab (or pembrolizumab) x3 cycles followed by IV nivolumab (or pembrolizumab) x3 cycles.
  Interventions: Drug: nivolumab; Drug: pembrolizumab
- IV to Subcutaneous (Active Comparator): IV nivolumab (or pembrolizumab) x3 cycles followed by SC nivolumab (or pembrolizumab) x3 cycles
  Interventions: Drug: nivolumab; Drug: pembrolizumab

INTERVENTIONS:
Drug: nivolumab — IV nivolumab (480mg Q4W), SC nivolumab (1200mg Q4W)
  Other Names: OPDIVO®
Drug: pembrolizumab — IV pembrolizumab (400mg Q6W) or SC pembrolizumab (790mg Q6W)
  Other Names: Keytruda®

SUMMARY:
The study will evaluate patient and Health Care Professional- reported preference for Subcutaneous (SC) compared with IV nivolumab administration or similarly for SC compared with IV pembrolizumab.

DETAILED DESCRIPTION:
The development of SC nivolumab and SC pembrolizumab was intended to provide patients, physicians and health care systems compelling advantages to reduce the burden associated with ICI administration. However, despite the results of CheckMate 76K, Hillman Cancer Center utilization of SC nivolumab is poor. This study aims to formally assess, from the patients' perspective, whether SC administration of ICI agents is preferable to IV administration. Key secondary objectives include physician experience with SC vs. IV administration, cancer-related efficacy endpoints, and safety. Patients who are pending initiation of nivolumab monotherapy or nivolumab-based chemotherapy or targeted therapy combinations (Cohort A-1) will be enrolled. However, patients who are already receiving nivolumab or other ICI but are willing to be switched to nivolumab monotherapy or nivolumab-based combinations may be eligible to enroll in a separate cohort (Cohort B-1). US FDA has accepted a Biologics License Application from Merck for SC pembrolizumab for an FDA action date of 9/23/2025. Should SC pembrolizumab achieve FDA approval, we will aim to open 2 separate cohorts to evaluate patient preference for SC vs. IV pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign a written informed consent document.
* Able to read and write in English.
* Must be eligible to receive nivolumab (Cohorts A-1, B-1) or pembrolizumab (Cohorts A-2, B-2) singly or in combination with other FDA-approved agents (TKIs or chemotherapy) according to standard of care practices, as determined by the clinical judgment of the investigator.
* Prior and concurrent therapy criteria

  o Patients should either be ICI-naïve (Cohorts A-1, A-2) or be currently receiving adjuvant or front-line PD-(L)1 based therapy singly or in combination with FDA-approved agents (TKIs or chemotherapy) (Cohorts B-1, B-2).
* Locally advanced or advanced/metastatic solid tumor for which nivolumab OR pembrolizumab is on-label.

  * NOTE: IV nivolumab is FDA-approved in the following indications: RCC, melanoma, NSCLC, SCCHN, UC, dMMR/MSI-H CRC, HCC, esophageal cancer, and gastric, gastroesophageal and esophageal adenocarcinoma (gastric/GEJ).
  * NOTE: IV pembrolizumab is FDA-approved in the following indications: RCC, melanoma, NSCLC, SCCHN, UC, dMMR/MSI-H CRC, HCC, esophageal cancer, gastric/GEJ, cervical cancer, cutaneous squamous cell carcinoma (cSCC), Merkel cell carcinoma (MCC), endometrial carcinoma, tumor mutational burden-high (TMB-H) cancers, triple negative breast cancer (TNBC).
* Cohort-specific criteria.

  * Cohort A-1: Patients who are treatment-naive (i.e. for whom nivolumab is planned but has not yet been initiated) are eligible to enroll.
  * Cohort B-1: Patients who are already receiving treatment with nivolumab (singly or in combination with TKI or chemotherapy) OR a different ICI-therapy but are willing to switch to nivolumab monotherapy or nivolumab based combinations may eligible to enroll if nivolumab is on-label for their cancer.
  * Cohort A-2: Patients who are treatment-naive (i.e. for whom pembrolizumab is planned but has not yet been initiated) are eligible to enroll.
  * Cohort B-2: Patients who are already receiving treatment with pembrolizumab (singly or in combination with TKI or chemotherapy) OR a different ICI-therapy but are willing to switch to pembrolizumab monotherapy or pembrolizumab based combinations may eligible to enroll if pembrolizumab is on-label for their cancer.
  * NOTE: Patients who are currently receiving nivolumab + ipilimumab combination as induction may be eligible to enroll in Cohort B-1 following induction (i.e. during planned maintenance) in indications including but not limited to advanced/metastatic melanoma, ccRCC, MSI-H/dMMR mCRC.
  * NOTE: Patients for whom nivolumab + ipilimumab combination is planned as maintenance are not eligible (i.e. NSCLC patients being treated per CheckMate-227 or CheckMate-9LA).
  * NOTE: Patients for whom anti-PD-1 based immunotherapy is planned as neoadjuvant therapy are not appropriate. Such patients may be considered for enrollment at the time of commencing adjuvant therapy in cohorts A-2 or B-2 as appropriate.

Exclusion Criteria:

* Participant unable to receive nivolumab (or pembrolizumab) due to prior allergic reactions to nivolumab (or pembrolizumab) or any of its ingredients.
* Has severe hypersensitivity (≥Grade 3) to nivolumab (or pembrolizumab) and/or any of its excipients.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Preference for Subcutaneous Nivolumab Treatment | Up to 48 months
  The proportion of patients with locally advanced or advanced/metastatic solid tumors who prefer SC to IV nivolumab.
Preference for Subcutaneous Pembrolizumab Treatment | Up to 48 months
  The proportion of patients with locally advanced or advanced/metastatic solid tumors who prefer SC to IV pembrolizumab.

SECONDARY OUTCOMES:
Therapy Administration Satisfaction Questionnaire | Up to 48 months
  Patient assessed satisfaction with SC vs. IV nivolumab (or pembrolizumab) using Therapy Administration Satisfaction Questionnaire (using TASQ-IV) in patients with locally advanced or advanced/metastatic solid tumors pending initiation of nivolumab (or pembrolizumab) monotherapy or nivolumab- (or pembrolizumab-) based combinations.
Therapy Administration Satisfaction Questionnaire | Up to 48 months
  Patient assessed satisfaction with SC vs. IV nivolumab (or pembrolizumab) using Therapy Administration Satisfaction Questionnaire (using TASQ-SC) in patients with locally advanced or advanced/metastatic solid tumors pending initiation of nivolumab (or pembrolizumab) monotherapy or nivolumab- (or pembrolizumab-) based combinations.
Health-Related Quality of Life (HRQoL) - EORTC QLQ-C30 | Screening Phase - Up to 28 days after signed consent
  Patient reported HRQoL scores using the EORTC QLQ-C30 instrument. The categories/domains include functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), global health status and quality of life scale. Item scoring for functional items is 1 (Not at all) to 4 (Very much); Item scoring for global health items is 1 (Very poor) to 7 (Excellent). Total scores (all items) range from 0 to 100. For functional and global quality of life scales higher scores mean a better level of functioning. For symptom-oriented scales, a higher score means more severe symptoms.
Health-Related Quality of Life (HRQoL) - EORTC QLQ-C30 | At Day 1 of Treatment Cycle 3
  Patient reported HRQoL scores using the EORTC QLQ-C30 instrument (30 items). The categories/domains include functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), and global health status and quality of life scale. Item scoring for functional and symptom items is 1 (Not at all) to 4 (Very much); Item scoring for global health items is 1 (Very poor) to 7 (Excellent). Total scores range from 0 to 100. For functional and global quality of life scales higher scores mean a better level of functioning. For symptom-oriented scales, a higher score means more severe symptoms.
Health-Related Quality of Life (HRQoL) - EORTC QLQ-C30 | At Day 1 of Treatment Cycle 6
  Patient reported HRQoL scores using the EORTC QLQ-C30 instrument (30 items). The categories/domains include functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), and global health status and quality of life scale. Item scoring for functional and symptom items is 1 (Not at all) to 4 (Very much); Item scoring for global health items is 1 (Very poor) to 7 (Excellent). Total scores range from 0 to 100. For functional and global quality of life scales higher scores mean a better level of functioning. For symptom-oriented scales, a higher score means more severe symptoms.
Change in Health-Related Quality of Life (HRQoL) - EORTC QLQ-C30 | Up to 48 nmonths
  Changes in patient reported HRQoL scores using the EORTC QLQ-C30 instrument. The categories/domains include functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), and global health status and quality of life scale. Item scoring for functional and symptom items is 1 (Not at all) to 4 (Very much); Item scoring for global health items is 1 (Very poor) to 7 (Excellent). Total scores range from 0 to 100. For functional and global quality of life scales higher scores mean a better level of functioning. For symptom-oriented scales, a higher score means more severe symptoms.
Health Related Quality of Life (HRQoL) - EQ-5D-5L | Screening Phase - Up to 28 days after signed consent
  Patient reported HRQoL scores using the EQ-5D-5L instrument. EQ-5D-5L is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from each of the five dimensions range from 1 to 5. Total score ranges from 5 to 25, where higher scores indicate worse health status.
Health Related Quality of Life (HRQoL) - EQ-5D-5L | At Day 1 of Treatment Cycle 3
  Patient reported HRQoL scores using the EQ-5D-5L instrument. EQ-5D-5L is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from each of the five dimensions range from 1 to 5. Total score ranges from 5 to 25, where higher scores indicate worse health status.
Health Related Quality of Life (HRQoL) - EQ-5D-5L | At Day 1 of Treatment Cycle 6
  Patient reported HRQoL scores using the EQ-5D-5L instrument. EQ-5D-5L is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from each of the five dimensions range from 1 to 5. Total score ranges from 5 to 25, where higher scores indicate worse health status.
Change Health Related Quality of Life (HRQoL) - EQ-5D-5L | Up to 48 months
  Change in patient reported HRQoL scores using the EQ-5D-5L instrument. EQ-5D-5L is a preference-based measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from each of the five dimensions range from 1 to 5. Total score ranges from 5 to 25, where higher scores indicate worse health status.
Physician-defined TTNT | Up to 48 months
  Physician-defined time to next therapy (TTNT) is defined as the period from the start of the treatment to the start of the next line of treatment.
Incidence of irAEs | Up to 48 months
  Incidence of immune-related adverse events (irAEs) that result in a dose hold or delay in patients treated with either SC or IV nivolumab (or pembrolizumab) per Common Terminology Criteria for Adverse Events (CTCAE) guidelines v5

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar J Davar, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No